CLINICAL TRIAL: NCT06719258
Title: Evaluation of Gas Humidification Practices in Patients Under Invasive Mechanical Ventilation: Benefit of the F & P950 Heated Humidifier: Comparison With the MR 850 on Clinical Events of Under-humidification
Brief Title: Evaluation of Gas Humidification Practices in Patients Under Invasive Mechanical Ventilation
Acronym: FP950
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal Investigator, Laval University
Other Study IDs: 2022-3714
Record Dates: First submitted 2024-11-20; First posted 2024-12-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Humidifier Lung; Mechanical Fragility; Respiratory Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MR850: 20 subjects on this heating humidifier (Fisher & Paykel MR850).
  Interventions: Device: MR850
- FP950: 20 subjects on this heating humidifier (Fisher & Paykel FP950).
  Interventions: Device: FP950

INTERVENTIONS:
Device: MR850 — This humidifier will be used straight away for patients whose intubation is expected to last longer than 24 hours.
  Groups: MR850
Device: FP950 — This humidifier will be used straight away for patients whose intubation is expected to last longer than 24 hours.
  Groups: FP950

SUMMARY:
When mechanical ventilation is initiated, a humidification method should be chosen. There is two methods: heat and humidity exchanger filters or heated humidity. The second method is recognized to be more efficient, but many external factors can influence its performance. Insufficient humidity results in observable problems, such as difficult management of respiratory secretions.

The study compare two heated humidifiers already used in ICU.

Data will be collected retrospectively from June 1, 2021.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Admitted to intensive care
* Under invasive mechanical ventilation with the usual indications for the use of a heated humidifier (prolonged invasive mechanical ventilation and / or protective ventilation requiring high respiratory rates.

Exclusion Criteria:

* Mechanical venitilation immediately after surgery (<24h)
* Imminent extubation or planned intubation of very short duration (<24h)
* Enrolled in the SAVE-ICU study in the group receiving volatile agents with the AnaConDa system.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient in ICU on ventilation will be consider.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Endotracheal tube occlusion requiring emergency tube change | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  Under-humidification episodes are defined as follows:
  - Occurence of endotracheal tube occlusion requiring emergency tube change
Bronchoscopy | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  Under-humidification episodes are defined as follows:
  - Occurence of performing a bronchoscopy for a suspected sub-occlusion (thick or sticky secretions), and the total number of bronchoscopies performed per patient
Tracheal saline instillations | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  Under-humidification episodes are defined as follows:
  - Occurence of tracheal saline instillations due to sticky secretions or suspected endotracheal tube sub-occlusion
Thick secretions | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  Under-humidification episodes are defined as follows:
  - Occurence of tracheal secretions describe at thick secretions (rated at 5 on the secretions scale used at the hospital) or "sticky secretions" if specified
Change humidifier settings | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  Under-humidification episodes are defined as follows:
  - The number of operations required to change humidifier settings if the plate temperature is below 62 degrees Celcius (with the MR850).

SECONDARY OUTCOMES:
Other elements that may be influenced by the quality of the humidification used during mechanical ventilation | At the end of the mechanical ventilation period or at 21 days ( the first of the 2 occurred)
  These data will be collected:
  * mechanical ventilation time
  * length of stay in intensive care
  * ventilation pressures
  * use of bronchodilator aerosols.
  * Ambien room air temperature

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec, Canada